CLINICAL TRIAL: NCT02423148
Title: A Pilot Study of a Novel Fluorescence Endoscopic Device for Sentinel Lymph Node Mapping in Lung Cancer in Combination With Indo-Cyanine Green
Brief Title: Pilot Study of Novel Fluorescence Endoscopic Device for Sentinel Lymph Node Mapping in Lung Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Co-investigator left facility. Decided not to enroll patients therefore.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Akorn, Inc. (Industry)
Responsible Party: Principal Investigator, Sidhu Gangadharan, Principal Investigators, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-441
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FluoSCOPE device (Experimental): All study interventions will occur intraoperatively during the subject's planned surgery. No deviation from standard of care will be performed with the exception of the following specific interventions:-
  * Intraoperative injection of indocyanine green (ICG) around tumor and imaging with the FluoSCOPE NIR endoscopic imaging system
  * Treatment will be administered on an inpatient basis
  Interventions: Drug: Indocyanine green (ICG); Device: FluoSCOPE

INTERVENTIONS:
Drug: Indocyanine green (ICG)
  Other Names: IC-Green
Device: FluoSCOPE

SUMMARY:
This research study is studying a new imaging method that will show lymph nodes in the lung during lung cancer surgery. The name of the study intervention involved in this study is:

-- The combination of the FluoSCOPE device and Indocyanine Green

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this study intervention. The FDA (the U.S. Food and Drug Administration) has not approved Indocyanine Green for your specific disease, but it has been approved for other uses.

In this research study, the investigators are interested in learning how a new investigational device, the FluoSCOPE, performs in the operating room. This study will also allow the investigators to optimize the settings of the imaging system. The investigators hope that this device, along with the local injection of Indocyanine Green around the tumor, will help find the sentinel lymph nodes in real-time during the surgery to remove lung cancer.

Although this is the first time the FluoSCOPE is being used in humans, the technology of near-infrared fluorescence imaging has been used for the detection of sentinel lymph nodes of patients with breast cancer, skin cancer and lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Participant must have histologically confirmed lung cancer and be deemed an appropriate surgical candidate for thoracoscopic lung resection and will have consent for a sentinel lymph node mapping by their oncologic surgeon. These patients will have invasive non-small cell lung cancers for which thoracoscopic mediastinal lymph node dissection at the time of thoracoscopic lung resection is standard of care. The extent of lung resections in potential trial patients could span from sublobar resection (i.e. wedge resection) to pneumonectomy, though it is anticipated that most patients will be undergoing the most common anatomic operation for lung cancer which is lobectomy.

All stages of lung cancer that would otherwise be undergoing thoracoscopic lung resection and mediastinal lymph node dissection would be eligible.

* Age minimum: 18 years.
* The minimum eligible subject age for this trial is 18 years. Individuals older than age 18 are typically cared for in adult oncology clinics at our institutions. Individuals under the age of 18 are excluded because safety studies including dosing or adverse event data in this population are currently not available. Essentially all of the patients operated upon for lung cancer at the BIDMC are adult men and women. Because of the nature of this disease, we do not anticipate, and will not be, enrolling any children into the study.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants who are receiving any other investigational agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to indocyanine green, including those patients with a history of iodide or seafood allergy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant or may become pregnant, as well as those women who are breastfeeding, will be excluded from this study. Pregnant women are excluded from this study because there is unknown risk associated with ICG (US FDA Risk Category C: there are no controlled studies in women, or no studies are available in either animals or women). Because there is an unknown, but potential, risk of adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated.
* Patients in whom the tumor might not be accessible for peritumoral injection of indocyanine green, e.g. small, central tumors.
* No other appropriate agent-specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11-03 (Actual); Study Completion 2016-11-03 (Actual)

PRIMARY OUTCOMES:
Sentinel lymph node(s) is identified via NIR fluorescence imaging | Day one

SECONDARY OUTCOMES:
Signal-to-background ratio | Day One
  signal-to-background ratio, determined by the relationship of field of view, fluence rate, and exposure time, is at least 2:1.
Number of Participants with Adverse Events | Day One

CONTACTS AND LOCATIONS:
Overall Officials: Sidhu Gangadharan, MD, Principal Investigator — Beth Israel Deaconess Medical Center